CLINICAL TRIAL: NCT05667129
Title: A Phase 1 Study to Evaluate Safety and Tolerability of Single and Multiple Ascending Doses of XEN-101
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xeno Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XB22-001
Record Dates: First submitted 2022-12-19; First posted 2022-12-28 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- XEN-101 (Experimental): Capsule formulation
  Interventions: Drug: XEN-101
- Placebo (Placebo Comparator): Capsule formulation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XEN-101 — Capsule formulation
  Arms: XEN-101
Drug: Placebo — capsule formulation
  Arms: Placebo

SUMMARY:
The goal of this study is to assess the safety and tolerability of single and multiple ascending doses of XEN-101

DETAILED DESCRIPTION:
Single ascending dose (SAD) study to evaluate the safety and tolerability of XEN-101 in healthy participants. Multiple ascending dose (MAD) study to evaluate the safety and tolerability of XEN-101 in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18-60 years at Screening
2. SAD part: BMI 18-30 kg/m2; MAD part 2a: BMI 22-27 kg/m2; MAD Part 2b: BMI 30-40 kg/m2
3. Stable body weight for at least 3 months (fluctuation of less than or equal to 5% and not exceeding 4 kg) in all study Parts.
4. Women of childbearing potential shall agree to use an adequate method of contraception from the date of signing of the informed consent, throughout the study, and for 4 weeks after the final (EOS) study visit. In addition, they must be advised not to donate ova during this period. From the date of signing of the informed consent, throughout the study, and for 8 weeks after the last dose of study medication, non sterilized male subjects who are sexually active with a female partner of childbearing potential must use barrier contraception (e.g., condom with spermicidal cream or jelly). In addition, they must be advised not to donate sperm during this period.
5. Females of childbearing potential must have a negative pregnancy test at Screening and on Day -1 (baseline)
6. Able to provide Informed Consent
7. Willing and able to comply with this protocol and procedures, including feces pro-cessing and be available for the entire duration of the study.

Exclusion Criteria:

1. Currently enrolled in another investigational device or drug study, or less than 30 days or 5 time the half-life of the drug candidate, whichever is longer, passed at Screening since ending the treatment period the previous investigational device or drug study
2. History of diabetes mellitus, hypertension, sleep apnea, liver, kidney, auto-immune disease
3. Current nicotine use or in past 6 months (smoking, vaping, etc)
4. Uncontrolled psychiatric disorder
5. History of eating disorder (e.g. anorexia nervosa, bulimia, binge-eating disorder)
6. History of alcohol, nicotine, or substance misuse in the last 5 years
7. Use of antibiotics, antivirals, antifungals during past 3 months
8. Use of proton pump inhibitors or non-stable dose antidepressants
9. Use of anti-obesity medications (e.g. GLP-analogues, stimulants, bupropri-on/naltrexone, etc.)
10. Use of obesogenic medications (e.g. anti-diabetics, anti-convulsives, anti-histamines, beta-blockers, etc.) in past 3 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
The frequency of adverse events (Safety of XEN-101) | From Day 1 through end of study (Day 7 SAD; Day 38 MAD)
  assessing the type and frequency of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Geza Lakner, MD, Principal Investigator — Clinical Research Units Hungary
Locations (1):
- CRU Hungary - Early Phase Unit, Kistarcsa, Hungary

IPD SHARING:
Plan to Share IPD: No